CLINICAL TRIAL: NCT04640935
Title: Retrospective Multicenter Study of Paclitaxel in Combination With Bevacizumab in Patients With Stage IV Non-small Cell Lung Cancer (NSCLC).
Brief Title: Paclitaxel in Combination With Bevacizumab in Patients With Stage IV NSCLC.
Acronym: AVATAX
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Annecy Genevois (Other)
Collaborators: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 19-09
Record Dates: First submitted 2020-11-09; First posted 2020-11-23 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non-small cell lung cancers; Paclitaxel; Bevacizumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to evaluate the paclitaxel-bevacizumab combination retrospectively and multicenter in current practice, with subgroup analyses of the following patients: patients who have previously received immunotherapy, patients with an EGFR or ALK oncogenic addiction pathway, patients who have previously received taxanes or anti-angiogenic agents.

DETAILED DESCRIPTION:
Lung and bronchopulmonary cancer is the leading cause of cancer death in France and worldwide. It is diagnosed at the metastatic stage from the outset in approximately 50% of cases. Non-small cell lung cancers (NSCLC) are the most frequent histological forms of lung cancer (approximately 85% of cases) with a predominance of the non-epidermal type.

The increase in the number of treatments available, improved supportive care and better patient selection have, in recent years, made it possible to expand the range of first-line chemotherapy treatments available at delà̀ and have contributed to the increase in overall survival (OS). As a result, nearly 80% of patients with metastatic NSCLC receive a second line of treatment. The main objective in these often symptomatic patients is a satisfactory tumor control rate with acceptable tolerability.

For a long time, the second-line reference chemotherapy has been docetaxel or pemetrexed as monotherapy with modest results. Alternative treatments such as the combination of paclitaxel (chemotherapy)-bevacizumab (anti-angiogenic monoclonal antibody) have been studied. Since 2010, by analogy with breast cancer and in the absence of therapeutic alternatives, the paclitaxel-bevacizumab doublet has been used in non-epidermal stage IV NSCLC in France. The value of combining taxane chemotherapy with an anti-angiogenic molecule has been demonstrated in two Phase 3 clinical trials. Thus, this combination is an integral part of the possible treatments in 2nd line and beyond, registered since 2016 in the treatment guidelines for non-epidermal NSCLC.

The first-line therapeutic strategy will also be redefined in 2019 with the use of immunotherapy for a majority of patients. Subsequent treatment lines will be modified, with a focus on chemotherapy, in particular the paclitaxel-bevacizumab combination.

As this combination has been used in current practice for several years, and in view of the upcoming changes to the first and second line of NSCLC treatment, data on the efficacy and tolerance of this combination in real life are needed to guide our practices. Recent studies are also looking at the efficacy of chemotherapy, particularly taxane chemotherapy associated with an anti-angiogenic agent after a previous line including immunotherapy, with a favorable signal.

The aim of the study is to evaluate the paclitaxel-bevacizumab combination retrospectively and multicenter in current practice, with subgroup analyses of the following patients: patients who have previously received immunotherapy, patients with an EGFR or ALK oncogenic addiction pathway, patients who have previously received taxanes or anti-angiogenic agents.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old;
* Histologically or cytologically confirmed diagnosis of non-epidermal NSCLC;
* Advanced stage IV disease at the start of treatment with paclitaxel-bevacizumab according to TNM 7/8th edition classification;
* Treatment with paclitaxel-bevacizumab received as second-line therapy or beyond, in a clinical trial or not;
* Alive patients not opposed to the use of their data

Exclusion Criteria:

* Patient under guardianship or curatorship at the date of the study ;
* Patients alive at the time of the study who are opposed to the use of their data
* Opposition to the use of their data expressed during the lifetime of patients who died at the time of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include all eligible patients who started paclitaxel-bevacizumab between January 1, 2010 and May 1, 2018. The number of patients is estimated to be approximately 200.
Sampling Method: Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2020-06-05 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | Up to 12 months
  Progression-free survival with paclitaxel-bevacizumab, i.e., the time from the start of paclitaxel-bevacizumab treatment to cancer progression, estimated at 12 months in the general population.

SECONDARY OUTCOMES:
Drugs administration dosage description | Up to 12 months
  Description of the different monthly drug administration regimens
Objective response rate and control rate | Up to 12 months
  Objective response rate and control rate according to RECIST 1.1 criteria in the general population
Overall survival Rate | Up to 12 months
  Overall survival, assessed on the whole population
Objective Response Rate | Up to 12 months
  Objective Response Rate in the following subgroups:
  * patients treated after immunotherapy and especially immediately after immunotherapy;
  * Patients with an oncogenic EGFR or ALK addiction pathway;
  * Patients previously treated with taxanes;
  * Patients previously treated with anti-angiogenic drugs;
Progression-Free Survival Rate | Up to 12 months
  Progression-Free Survival in the following subgroups:
  * patients treated after immunotherapy and especially immediately after immunotherapy;
  * Patients with an oncogenic EGFR or ALK addiction pathway;
  * Patients previously treated with taxanes;
  * Patients previously treated with anti-angiogenic drugs;
Disease Control Rate | Up to 12 months
  Disease Control in the following subgroups:
  * patients treated after immunotherapy and especially immediately after immunotherapy;
  * Patients with an oncogenic EGFR or ALK addiction pathway;
  * Patients previously treated with taxanes;
  * Patients previously treated with anti-angiogenic drugs;
Overall Survival Rate | Up to 12 months
  Overall Survival in the following subgroups:
  * Patients treated after immunotherapy and especially immediately after immunotherapy;
  * Patients with an oncogenic EGFR or ALK addiction pathway;
  * Patients previously treated with taxanes;
  * Patients previously treated with anti-angiogenic drugs;
Frequency of safety events | Up to 12 months
  Frequency of grade ≥3 adverse events and frequency of discontinuation of paclitaxel-bevacizumab for toxicity ;

CONTACTS AND LOCATIONS:
Overall Officials: Chantal Decroisette, Principal Investigator — CH Annecy Genevois
Locations (15):
- France (15):
  - Hôpital Ambroise Paré AP-HP, Boulogne-Billancourt
  - Centre Hospitalier Universitaire Brest, Brest
  - Centre Hospitalier Métropole Savoie, Chambéry
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Centre Hospitalier Universitaire Grenoble Alpes, Grenoble
  - Centre Hospitalier de Versailles André Mignot, Le Chesnay
  - Centre Hospitalier Universitaire de Lille, Lille
  - Centre Léon Bérard Lyon, Lyon
  - Hospices Civils de Lyon, Lyon
  - Centre Hospitalier François Quesnay, Mantes-la-Jolie
  - Centre Hospitalier Annecy Genevois, Metz-Tessy
  - Institut Curie, Paris
  - Institut Curie Saint Cloud, Saint-Cloud
  - Institut de Cancérologie Lucien Neuwirth, Saint-Etienne
  - Hôpital Foch, Suresnes